CLINICAL TRIAL: NCT01196312
Title: Novel Intervention for Drug Use and HIV Risk Among Anxiety Sensitive Heroin Users
Brief Title: Anxiety Sensitivity Treatment for Heroin Users
Acronym: ASTH-HR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Joe Smith, Director - HRPP (C. Lejuez is no longer at UMD), University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA023384
Record Dates: First submitted 2010-08-23; First posted 2010-09-08 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Anxiety
Keywords: anxiety sensitivity; heroin
MeSH Terms: conditions — Anxiety Disorders

INTERVENTIONS:
Behavioral: Anxiety sensitivity therapy — ASTH consists of 6 sessions of individual treatment, each lasting approximately 75 minutes over 3 weeks. In general, each session consists of the following components1) psychoeducation regarding the anxiety response, with a focus on increasing awareness of the ways in which the patient interprets or evaluates that response 2) assistance in developing healthy emotion regulation strategies that can be used to increase acceptance and tolerance of the anxiety response (including associated catastrophic thoughts), as well as understanding the consequences associated with avoidance or control of anxiety 3) a minimum of 3 interoceptive exercises tailored to activate feared anxiety-related sensations and 4) daily homework assignments (i.e., daily anxiety monitoring and interoceptive exercises).

SUMMARY:
Anxiety Sensitivity Treatment for Heroin Users is a development project targeting mild and above levels of anxiety sensitivity that will involve the testing of a specialized protocol for improving treatment retention and outcomes for heroin dependent individuals in a residential substance use treatment. ASTH-HR will integrate established treatment modules such as Healthy Relationships, along with interoceptive exposure, affect management, and psycho-education exercises developed for anxiety prevention and treatment programs with standard substance use treatment.

ELIGIBILITY:
Inclusion Criteria:

* exhibit a score of 21 on a self-report measure of anxiety sensitivity
* be in 28 days of residential substance use treatment.
* meet criteria for current opioid dependence as determined by SCID interview administered at intake.

Exclusion Criteria:

* evidence of limited mental competency
* the inability to give informed, voluntary, written consent to participate
* current psychosis
* current bipolar disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 | 24 weeks

SECONDARY OUTCOMES:
Timeline Follow Back 90 days | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Salvation Army Harbor Light Treatment Facilitiy, Washington D.C., District of Columbia, United States